CLINICAL TRIAL: NCT06059235
Title: Concordance : a New Concept for Clinical Pharmacy in Partnership With Patients at a Geriatric Day Clinic
Acronym: COPAPI-G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COPAPI-G
Record Dates: First submitted 2023-03-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adherence, Medication
Keywords: pharmaceutical care; geriatrics; consultation; medication review
MeSH Terms: conditions — Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Package of clinical pharmacy activities including :
  * Medication history (during assessment consultation)
  * Medication review and consultation with the geriatrician
  * Therapeutic education (during results consultation)
  * Shared decision (at results consultation)
  * One-week follow-up call + usual care
  Interventions: Other: pharmaceutical care
- controle (No Intervention): Medication history (during assessment consultation) + usual care

INTERVENTIONS:
Other: pharmaceutical care — consultation with a pharmacist performing advanced pharmaceutical care : Package of clinical pharmacy activities including :
  Medication history (during assessment consultation) Medication review and consultation with the geriatrician Therapeutic education (during results consultation) Shared decision (at results consultation) One-week follow-up call + usual care
  Arms: intervention

SUMMARY:
The goal of this clinical trial is to assess the impact of pharmaceutical consultations in older patients having a comprehensive geriatric assessment at geriatric day-clinic. The main question it aims to answer is: What is the impact on patient adherence Participants will benefit from medication history taking, medication review, therapeutic education, shared decision-making and follow-up phone call. Researchers will compare with a control group, benefiting from medication history taking and usual care from the geriatric day-clinic.

DETAILED DESCRIPTION:
Research question: What is the impact of a clinical pharmacy activity (including a medication history, a medication review, therapeutic education, a shared decision step and a follow-up call) on medication adherence in elderly patients followed up for geriatric assessment at the geriatric day hospital? Design: Intervention study, randomized, controlled, open-label, with evaluation at 2 months. The study will run from January 1, 2023 to September 1, 2024 (20 months), at the CUSL geriatric day hospital.

Participants: patients admitted to the geriatric day hospital for a geriatric assessment will be eligible for the project. A geriatric assessment comprises 2 consultations at the geriatric day hospital: a "assessment" consultation, where the patient meets the members of the multidisciplinary team, and a "results" consultation, where the geriatrician provides the patient with care recommendations.

The general practitioners, pharmacists and nursing home referral nurse (if applicable) of the participants in the intervention group will be invited to take part in a satisfaction survey.

Intervention: The intervention includes several clinical pharmacy activities

* Medication history (during assessment consultation)
* Medication review and consultation with the geriatrician
* Therapeutic education (during results consultation)
* Shared decision-making (during results consultation)
* One-week follow-up call Control: usual care. Outcomes: primary: comparison at 1.5 months (telephone FUP) after outcome consultation of ASK-20 total Adherence Survey score (measures medication adherence and identifies barriers to adherence).

Secondary outcomes measured at 1.5 months:

* ASK-20 TBC measures
* EQ5D quality-of-life scores
* number of inappropriate medications according to STOPP&START
* number of drug interactions DDI
* pain score
* hospital admissions during the FUP period Various indicators related to pharmaceutical activity will also be collected.

This project will serve as a rationale for the long-term development of a clinical pharmacy activity at the day hospital, and will help maintain CUSL's status as an innovator in clinical pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* 75+
* patients admitted to the geriatric day hospital for a geriatric assessment will be eligible for the project. A geriatric assessment comprises 2 consultations at the geriatric day hospital: a "major assessment" consultation, where the patient meets the members of the multidisciplinary team, and a "results" consultation, where the geriatrician provides the patient with care recommendations.

Exclusion Criteria:

* less than 75
* not speaking French
* exlusion based on geriatrician advice

Ages: 75 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
presence of barriers to adherence as measured by ASK-20 score (the sum of raw ASK-20 item scores) | 6weeks
  ASK-20 (questionnaire) consists of 20 clinically actionable items representing multiple factors that affect medication adherence. Each of the 20 items score from 1 to 5. A score of 20 means low barriers to adherence; A score of 100 means maximum barriers to adherence. Comparizon of ASK-20 score from baseline to 6weeks in both arms. Hahn SR, Park J, Skinner EP, Yu-Isenberg KS, Weaver MB, Crawford B, Flowers PW. Development of the ASK-20 adherence barrier survey. Curr Med Res Opin. 2008 Jul;24(7):2127-38. doi: 10.1185/03007990802174769. Epub 2008 Jun 12. PMID: 18554431.

SECONDARY OUTCOMES:
count of barriers to adherence measured by TBC ASK-20 (Total Barrier Count) | 6weeks
  Each of the 20 items Of the ASK-20 (questionnaire) was dichotomized as positive - indicating a barrier, or negative. TBC counts the barriers per patient. Comparison of TBC from baseline to 6 weeks in both arms. Hahn SR, Park J, Skinner EP, Yu-Isenberg KS, Weaver MB, Crawford B, Flowers PW. Development of the ASK-20 adherence barrier survey. Curr Med Res Opin. 2008 Jul;24(7):2127-38. doi: 10.1185/03007990802174769. Epub 2008 Jun 12. PMID: 18554431.
quality of life measured with EQ5D (Visual analogical scale) score | 6weeks
  Quality of life questionnaire. Comparison of estimated quality of life between baseline and 6 weeks in both arms
number of inappropriate medications per patient according to STOPP/START | 6weeks
  Detection od potentially inappropriate medications (PIM) using STOPP&START version 2 in medication treatment and comparison of number of PIM between baseline and 6 weeks in both arms
number of Drug-drug interactions per patient from the Anrys list | 6weeks
  Comparison in both arms of drug-drug interactions detected at baseline and 6 weeks in medication treatment according to Anrys et al. Anrys P, Spinewine A. An International Consensus List of Potentially Clinically Significant Drug-Drug Interactions in Older People: Clinical Utility? J Am Med Dir Assoc. 2022 Mar;23(3):522. doi: 10.1016/j.jamda.2021.11.038. Epub 2022 Jan 10. PMID: 35026145.
pain severity (from EQ-D) | 6weeks
  Comparison of pain reported in EQ5D questionnaire from baseline to 6 weeks in both groups
number of hospital admissions reported by patient | 6weeks
  comparison of reported hospitalisations in both groups during the study period (questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No